CLINICAL TRIAL: NCT03728725
Title: Multicentre Clinical Trial to Assess the Performance of the Xpert MTB/XDR Assay for INH- and Second-line Resistance Detection
Brief Title: Xpert MTB/XDR Clinical Evaluation Trial
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Cepheid (Industry); PD Hinduja Hospital and Medical Research Centre, Mumbai, India (Unknown); Phthisiopneumology Institute, Chisinau, Moldova (Unknown); National Institute of Tuberculosis and Respiratory Disease, New Delhi, India (Unknown); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: 7162-02/2
Record Dates: First submitted 2018-10-05; First posted 2018-11-02 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2020-04

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum will be collected from consenting, enrolled adult participants. Sputum samples may voluntarily be stored for up to 20 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TB case detection Group: Patients with pulmonary TB symptoms and at least one DR-TB risk factor will be screened by Xpert MTB/RIF or Ultra. Patients with a clear TB-positive and RIF-resistant or RIF-sensitive result by Xpert MTB/RIF or Ultra and who consent to study procedures will be tested by Xpert MTB/XDR.
  Interventions: Device: Cepheid Gene Xpert MTB/XDR
- RIF-resistance MTB Group: An anticipated 316 additional RIF-resistant patients, as detected by Xpert MTB.
  /RIF, will be enrolled in this study to evaluate sensitivity and specificity of the Xpert MTB/XDR test against strains with other potential drug-resistance mutations.
  Interventions: Device: Cepheid Gene Xpert MTB/XDR

INTERVENTIONS:
Device: Cepheid Gene Xpert MTB/XDR — The Xpert MTB/RIF assay (Cepheid, Sunnyvale, CA) is an integrated, automated, cartridge-based system for MDR-TB diagnosis that uses the GeneXpert instrument platform. WHO confirmed evidence to support the widespread use of the Xpert MTB/RIF assay in 2010 and the assay has since been widely used in TB programs, but it is only capable of identifying Mycobacterium tuberculosis (Mtb) and detecting RIF resistance. The Xpert MTB/XDR assay will be evaluated for INH and second-line resistance detection, and to recommend its use in diverse clinical settings. The focus of this protocol is the multicentre clinical evaluation.

SUMMARY:
FIND and partners intend to address the need for a multi- and extensively drug-resistant tuberculosis (M/XDR-TB) diagnostic solution for patients in settings with a high burden of drug-resistant tuberculosis (DR-TB) though the development, evaluation and introduction of an Xpert MTB/XDR assay

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 years or above;

  * Symptoms suggesting pulmonary TB, i.e. persistent cough (generally ≥3 weeks or as per local definition of TB suspect), and at least one of the following:

    * Previously received >1 month of treatment for a prior TB episode or
    * Failing TB treatment with positive sputum smear or culture after ≥3 months of a standard TB treatment or
    * Had close contact with a known drug-resistant TB case or
    * Newly diagnosed with MDR-TB within the last 30 days or
    * Previously diagnosed with MDR-TB and failed TB treatment with positive sputum smear or culture after ≥3 months of a standard MDR-TB treatment regimen

Patients meeting the above criteria will be screened by Xpert MTB/RIF or Xpert MTB/RIF Ultra. TB patients meeting the following criteria will be included in the study:

* A clear Mtb-positive and RIF-resistant or RIF-sensitive result by Xpert MTB/RIF or Xpert MTB/RIF Ultra
* Provision of informed consent;
* Production of an adequate quantity (>3mL) of sputum

Exclusion Criteria:

* Participants will be excluded from the study if informed consent is not provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who have one or more risk factors for DR-TB presenting to participating centres will be screened by Xpert MTB/RIF or Ultra. Those who test MTB-positive by Xpert MTB/RIF or Ultra at the study sites will be asked to participate. Individuals will be recruited at outpatient clinic settings and inpatient hospital settings. HIV-positive individuals and HIV-negative individuals will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Estimate the diagnostic accuracy of the Xpert MTB/XDR assay for INH and ETH resistance detection | Day 1
  Sensitivity and specificity estimates for INH and ETH resistance detection
Estimate the diagnostic accuracy of the Xpert MTB/XDR assay for fluoroquinolone resistance detection | Day 1
  Sensitivity and specificity estimates for fluoroquinolone resistance detection
Estimate the diagnostic accuracy of the Xpert MTB/XDR assay for second-line injectable resistance detection | Day 1
  Sensitivity and specificity estimates for second-line injectable resistance detection

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Pthisiopenumology, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: Yes
Data sharing statement Individual, de-identified participant data will be shared, including data dictionaries. Other documents that have been made available include the study protocol and statistical analysis plan. Templates of the informed consent forms may be shared upon request. The data will be available immediately following publication with no end date. The data will be shared with anyone who wishes to access the data. The data will be available for any purpose of analyses. For data, please contact the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon publication of final study results
Access Criteria: The data will be shared with anyone who wishes to access the data.

REFERENCES:
- [Derived] Penn-Nicholson A, Georghiou SB, Ciobanu N, Kazi M, Bhalla M, David A, Conradie F, Ruhwald M, Crudu V, Rodrigues C, Myneedu VP, Scott L, Denkinger CM, Schumacher SG; Xpert XDR Trial Consortium. Detection of isoniazid, fluoroquinolone, ethionamide, amikacin, kanamycin, and capreomycin resistance by the Xpert MTB/XDR assay: a cross-sectional multicentre diagnostic accuracy study. Lancet Infect Dis. 2022 Feb;22(2):242-249. doi: 10.1016/S1473-3099(21)00452-7. Epub 2021 Oct 7. PMID 34627496

DOCUMENTS (2):
  • Study Protocol (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03728725/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT03728725/SAP_001.pdf